CLINICAL TRIAL: NCT04768530
Title: Nitazoxanide as a New Local Adjunctive to Nonsurgical Treatment of Moderate Periodontitis: Clinical and Biochemical Evaluation
Brief Title: Nitazoxanide as a New Local Adjunctive to Nonsurgical Treatment of Moderate Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maha Talaab (Other)
Responsible Party: Sponsor-Investigator, Maha Talaab, Associate Professor, Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology department, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Nitazoxanide & periodontitis
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scaling and Root Planing (SRP) (Active Comparator)
  Interventions: Procedure: Scaling and Root Planing
- Scaling and Root Planing with Nitazoxanide hydrogel (Experimental)
  Interventions: Drug: Nitazoxanide hydrogel

INTERVENTIONS:
Procedure: Scaling and Root Planing — Supra- and sub-gingival calculus and debris were removed
  Arms: Scaling and Root Planing (SRP)
Drug: Nitazoxanide hydrogel — Scaling and root planing was performed in combination with the subgingivally delivered thermosensitive Nitazoxanide hydrogel as adjunct antimicrobial therapy.
  Arms: Scaling and Root Planing with Nitazoxanide hydrogel

SUMMARY:
The aim of the study was to assess the effect of nitazoxanide delivered subgingivally as thermosensitive hydrogel on the clinical and biochemical outcomes of SRP in patients with moderate periodontitis.

DETAILED DESCRIPTION:
A randomized, controlled clinical trial in a split-mouth design was conducted on forty patients equally divided between two groups: a control group treated with full mouth scaling and root planing (SRP) and a test group treated with SRP combined with subgingivally delivered 0.01% NTZ sustained release Poloxamer 407/hyaluronic acid thermosensitive hydrogel.

ELIGIBILITY:
Inclusion Criteria:

* Patients having probing depth (PD) ≥5 mm.
* Patients having bleeding on probing (BOP) in proximal tooth surface.
* Patients who could maintain an O'Leary plaque index ≤10 proceeded into the study.

Exclusion Criteria:

* Patients having any systemic disease that may affect the treatment outcomes.
* Smokers.
* Pregnant females.
* Patients receiving contraindicated medications, chemotherapy, or radiotherapy in the previous year.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Probing depth | up to 6 months
  Probing depth was recorded at tested sites with graduated William's probe graduated in 1 mm increment. Readings were rounded to the nearest mm.
Clinical attachment loss | up to 6 months
  Clinical attachment loss was recorded at tested sites with graduated William's probe graduated in 1 mm increment. Readings were rounded to the nearest mm.
Bleeding on probing | up to 6 months
  Bleeding on probing was assessed at tested sites with graduated William's probe graduated in 1 mm increment, within 15 seconds after probing, using a dichotomous scoring system (+ and -) for presence or absence, respectively.
Gingival index | up to 6 months
  Gingival index was assessed at 4 sites on six index teeth. Scores range from 0 to 3, with 0 being normal and 3 being severe inflammation
Biochemical assessment of inflammation | up to 6 months
  This involved determination of the gingival crevicular fluid (GCF) levels of matrix metalloproteinase 8 (MPP-8). A GCF sample was taken from the area showing the deepest pocket depth around the treated area.The samples were diluted in phosphate buffer saline (PBS) up to 1 mL. After waiting for 15 min, the paper points were removed, and 500 μL were centrifuged at 400 g for 4 min, then frozen at -20°C pending MMP-8 analysis using Human Matrix metalloproteinase 8/Neutrophil collagenase (MMP-8) ELISA Kit according to the manufacturer instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Maha R. Taalab, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Sylvia Farid, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Shaimaa Maklad, PhD, Study Director — Department of Pharmaceutics, Faculty of Pharmacy, Alexandria University, Egypt; Labiba El-Khordagui, PhD, Study Director — Department of Pharmaceutics, Faculty of Pharmacy, Alexandria University, Egypt; Maha El Tantawi, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt